CLINICAL TRIAL: NCT00017303
Title: A Phase II Trial Of IM862 Combined With Paclitaxel And Carboplatin In Newly Diagnosed Advanced Epithelial Ovarian Or Primary Peritoneal Carcinoma Followed By IM862 Consolidation Therapy
Brief Title: Combination Chemotherapy Plus IM-862 in Treating Patients With Resected Stage III Ovarian Cancer or Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cytran (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068674; CYTRAN-IM862-302; FHCRC-5156
Record Dates: First submitted 2001-06-06; First posted 2004-02-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2002-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: oglufanide disodium
Drug: paclitaxel
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. IM-862 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill tumor cells. Combining chemotherapy and IM-862 may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combination chemotherapy and IM-862 in treating patients who have resected stage III ovarian cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete pathologic response rate at second-look surgery in patients with optimally resected stage III ovarian epithelial or primary peritoneal cancer treated with adjuvant paclitaxel, carboplatin, and IM-862. II. Determine the safety profile of this regimen in this patient population. III. Determine the incidence of infectious and hematologic complications in patients treated with this regimen. IV. Determine the progression-free survival of patients with no disease or minimal disease burden after initial therapy, when treated with IM-862 consolidation therapy. V. Correlate angiogenesis markers and immunologic parameters with response in patients treated with this regimen.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to participating center. Patients are randomized to one of three IM-862 doses. Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Treatment with IM-862 begins within 10 days of chemotherapy initiation and continues until clinical evidence of disease progression or until 3 days before second-look surgery. Arm I: Patients receive a low-dose of IM-862 and 2 placebo doses intranasally daily. Arm II: Patients receive a medium-dose of IM-862 and 2 placebo doses as in arm I. Arm III: Patients receive higher-dose IM-862 intranasally three times daily. Patients undergo second-look surgery within 4-8 weeks after completion of the last course of chemotherapy. Patients with a complete pathologic response or only microscopically detectable residual disease receive consolidation therapy with IM-862, according to their original treatment arm. Consolidation therapy begins within 3-14 days after second-look surgery and continues for 24 weeks in the absence of disease progression. Patients are followed at 6 and 12 months.

PROJECTED ACCRUAL: A total of 180 patients (60 per arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III ovarian epithelial cancer or primary peritoneal carcinoma of one of the following cell types: Serous adenocarcinoma Mucinous adenocarcinoma Clear-cell adenocarcinoma Endometrioid Adenocarcinoma (not otherwise specified) Undifferentiated carcinoma Transitional cell Malignant Brenner's tumor Mixed epithelial carcinoma No borderline tumor (tumor of low malignant potential) Underwent prior standard initial cytoreductive surgery within the past 6 weeks Optimally resected disease with no residual site of disease more than 1 cm in greatest dimension Removal of all disease extending beyond the reproductive tract Total hysterectomy and bilateral salpingo-oopherectomy at cytoreductive surgery or in the past

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN SGOT no greater than 3 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix or breast No other major systemic medical illness that would preclude survival No poor general condition or medical, social, or psychosocial factors that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy for current malignancy At least 5 years since prior gene therapy At least 1 year since prior interleukin-2 (IL-2) At least 1 year since prior sargramostim (GM-CSF) Concurrent filgrastim (G-CSF) allowed No concurrent gene therapy No concurrent GM-CSF No concurrent IL-2 No other concurrent angiogenesis inhibitors (e.g., thalidomide, cyclooxygenase-2 inhibitors (e.g., rofecoxib or celecoxib), interferon products, or angiotensin-converting enzyme inhibitors) Chemotherapy: At least 5 years since prior anticancer chemotherapy No prior chemotherapy for current malignancy No other concurrent chemotherapy Endocrine therapy: No prior endocrine therapy for current malignancy At least 1 year since prior tamoxifen No concurrent tamoxifen Radiotherapy: No prior radiotherapy for current malignancy Surgery: See Disease Characteristics Other: At least 1 year since prior experimental or investigational medications No other concurrent experimental or investigational medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Paley, MD, Study Chair — Pacific Gynecology Specialists
Locations (19):
- United States (19):
  - Comprehensive Cancer Center, Glendale, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Stanford University Medical Center, Stanford, California
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Kansas School of Medicine-Wichita, Wichita, Kansas
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center - Las Vegas, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961